CLINICAL TRIAL: NCT05086848
Title: A Phase Ib Study to Evaluate Tolerability, Safety and Pharmacokinetics of Irinotecan Hydrochloride Liposome Injection in Combination With 5-FU/LV in Patients With Advanced Solid Tumors
Brief Title: A Study of Irinotecan Hydrochloride Liposome in Combination With 5-FU/LV in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YLTKL-Ib
Record Dates: First submitted 2021-09-29; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: a dose-escalation and expansion study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group: (Experimental): Irinotecan liposome plus 5-fluorouracil, Leucovorin
  Interventions: Drug: Irinotecan liposome、5-fluorouracil、Leucovorin

INTERVENTIONS:
Drug: Irinotecan liposome、5-fluorouracil、Leucovorin — Irinotecan liposome、5-fluorouracil、Leucovorin

SUMMARY:
This is a dose-escalation and expansion, open label, single centre, phase Ib study. In this study, the tolerability, safety, pharmacokinetics and efficacy of irinotecan hydrochloride liposome injection in combination with 5-FU/LV were studied in patients with advanced solid tumors. Meanwhile, to determine the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of irinotecan hydrochloride liposome.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid tumors documented as advanced or metastatic disease;
2. Subjects must be considered relapsed or refractory to standard therapies, have been intolerant to standard therapies, or have refused standard therapy;
3. ECOG: 0-1;
4. Adequate organ and bone marrow function;
5. sign an informed consent.

Exclusion Criteria:

1. Patients with brain malignant tumor or active CNS metastasis;
2. UGT1A1*28 homozygous mutants;
3. Clinically significant GI disorders;
4. Significant cardiovascular disease;
5. Active infection or uncontrolled fever;
6. Pregnant or breast feeding patients;
7. Allergic to a drug ingredient or component;
8. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Adverse Event (AE) | Assessed from study inclusion to 30 days after last dose
  Assessed by CTCAE v4.03
Dose Limiting Toxicities (DLT) | DLTs will be evaluated during 28-day period following the first dose of study treatment
  Dose Limiting Toxicities for patients in combination treatment
Maximal tolerated dose (MTD) | after the last patient in each cohort up to 12 months
  Maximum tolerated dose for patients in combination treatment

SECONDARY OUTCOMES:
Objective Response Rate | maximum time on study 12 months
  Objective response rate was based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
Progression Free Survival | The maximum time in follow up was 12 months
  Progression-free survival was defined as the time from the date of randomization to the date of disease progression, or death (any cause) on or prior to the clinical cutoff date, whichever occurs first.
Time to reach maximum plasma concentration (Tmax) | up to 168 hours after the first dose
  Tmax of total irinotecan, free irinotecan and SN-38
Maximum observed plasma concentration (Cmax) | up to 168 hours after the first dose
  Cmax of total irinotecan, free irinotecan and SN-38
Area under the plasma concentration versus time curve from time zero to time of last observed concentration (AUC0-t) | up to 168 hours after the first dose
  AUC0-t of total irinotecan, free irinotecan and SN-38
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-inf) | up to 168 hours after the first dose
  AUC0-inf of total irinotecan, free irinotecan and SN-38
Elimination half-life (T1/2) | up to 168 hours after the first dose
  T1/2 of total irinotecan, free irinotecan and SN-38
Clearance of drug from plasma (CL) | up to 168 hours after the first dose
  CL of total irinotecan
Volume of distribution (Vss) | up to 168 hours after the first dose
  Vss of total irinotecan

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ji D, Shen W, Li T, Wang H, Bai J, Cao J, Hu X. Liposomal irinotecan (HR070803) in combination with 5-fluorouracil and leucovorin in patients with advanced solid tumors: a phase 1b dose-escalation and expansion study. Invest New Drugs. 2024 Aug;42(4):462-470. doi: 10.1007/s10637-024-01442-2. Epub 2024 Jul 22. PMID 39037543